CLINICAL TRIAL: NCT00393198
Title: Multicenter Study to Investigate the Bleeding Profile and the Insertion Easiness in Women Inserted With a Second Consecutive MIRENA for Contraception or Menorrhagia
Brief Title: Bleeding Pattern and User Satisfaction During Second Consecutive MIRENA® in Contraception and Treatment of Menorrhagia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91473; 2006-000394-30 (EudraCT Number); 309988 (Other: Company internal)
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Contraception; Menorrhagia
Keywords: Intrauterine System; Contraception; Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Levonorgestrel (Mirena, BAY86-5028)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Cytotec
- Arm 3 (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levonorgestrel (Mirena, BAY86-5028) — Removal of first MIRENA and insertion of the second MIRENA at entry visit. Removal of MIRENA (in vitro release rate 20 microgram/24h) at year 5 visit.
  Arms: Arm 1
Drug: Cytotec — Cytotec, single, sublingual dose of 400 microgram, 3 hours prior to the MIRENA removal and insertion procedure at entry visit
  Arms: Arm 2
Drug: Placebo — Placebo, single, sublingual dose, 3 hours prior to the MIRENA removal and insertion procedure at entry visit.
  Arms: Arm 3

SUMMARY:
The purpose of this study is to assess the bleeding pattern during the last 3 months of the first MIRENA® and the first year of the second MIRENA® use.

DETAILED DESCRIPTION:
This study has previously been posted by Schering AG, Germany. Schering AG has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Woman currently using MIRENA for contraception or menorrhagia with duration use between 4 years 3 months and 4 years 9 months and willingness to continue with the method.
* Normal size uterus at insertion, corresponding to sound measure of 6-10 cm.
* Clinically normal cervical smear result within 12 preceding months or at screening.
* Clinically normal breast examination findings. For patients >/= 40 years at screening, a clinically normal mammography result within 12 preceding months or at screening is required.

Exclusion Criteria:

* Menopausal symptoms impairing patient's quality of life or current estrogen therapy for menopausal symptoms.
* Known or suspected pregnancy.
* Any distortion of the uterine cavity, including congenital or acquired uterine anomalies and fibroids distorting the uterine cavity.
* Current or recurrent pelvic inflammatory disease.
* Abnormal uterine bleeding of unknown origin.
* Acute cervicitis or vaginitis not responding to treatment.
* History of, diagnosed or suspected genital or other malignancy (excluding treated squamous cell carcinoma of the skin), and untreated cervical dysplasia.
* Any active acute liver disease or liver tumor.

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2006-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variable will be bleeding profile | Screening, entry (60-90 days after screening), month 3 and 6, year 1,2,3,4 and 5

SECONDARY OUTCOMES:
Secondary efficacy variables will be insertion assessment, continuation rate, pregnancy rate and menstrual comfort and user satisfaction | Screening, entry (60-90 days after screening), month 3 and 6, year 1,2,3,4 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Finland (6):
  - Helsinki
  - Hyvinkää
  - Jyväskylä
  - Kuopio
  - Tampere
  - Turku
- France (6):
  - Brignoles
  - Compiègne
  - Nancy
  - Quetigny
  - Reims
  - Roanne
- Ireland (2):
  - Mallow, Cork
  - Drogheda
- Stockholm, Sweden

REFERENCES:
- [Result] Heikinheimo O, Inki P, Kunz M, Parmhed S, Anttila AM, Olsson SE, Hurskainen R, Gemzell-Danielsson K. Double-blind, randomized, placebo-controlled study on the effect of misoprostol on ease of consecutive insertion of the levonorgestrel-releasing intrauterine system. Contraception. 2010 Jun;81(6):481-6. doi: 10.1016/j.contraception.2010.01.020. Epub 2010 Mar 1. PMID 20472114
- [Result] Gemzell-Danielsson K, Inki P, Boubli L, O'Flynn M, Kunz M, Heikinheimo O. Bleeding pattern and safety of consecutive use of the levonorgestrel-releasing intrauterine system (LNG-IUS)--a multicentre prospective study. Hum Reprod. 2010 Feb;25(2):354-9. doi: 10.1093/humrep/dep426. Epub 2009 Dec 1. PMID 19955104
- [Result] Heikinheimo O, Inki P, Kunz M, Gemzell-Danielsson K. Predictors of bleeding and user satisfaction during consecutive use of the levonorgestrel-releasing intrauterine system. Hum Reprod. 2010 Jun;25(6):1423-7. doi: 10.1093/humrep/deq079. Epub 2010 Apr 8. PMID 20378611
- [Derived] Heikinheimo O, Inki P, Schmelter T, Gemzell-Danielsson K. Bleeding pattern and user satisfaction in second consecutive levonorgestrel-releasing intrauterine system users: results of a prospective 5-year study. Hum Reprod. 2014 Jun;29(6):1182-8. doi: 10.1093/humrep/deu063. Epub 2014 Mar 28. PMID 24682613